CLINICAL TRIAL: NCT04487470
Title: Impact of Cigar Flavor on Tobacco Use Behaviors and Addiction in Dual Users
Brief Title: Impact of Cigar Flavor in Dual Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Erin Mead-Morse, Assistant Professor, UConn Health
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 19-202-2; K01DA048494 (NIH)
Record Dates: First submitted 2020-07-14; First posted 2020-07-27 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Tobacco Use Disorder
Keywords: Dual Tobacco Use; Smoking; Cigar Smoking; Cigarette Smoking
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Cigar Smoking; Cigarette Smoking

STUDY DESIGN:
Intervention Model Description: Randomized cross-over study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flavored Filtered Cigars (Experimental): Half of the group will be randomized to start with flavored filtered cigars (FCs) at the second visit and cross over to unflavored FCs at the third visit. FCs will be Cheyenne filtered cigars.
  Interventions: Other: Flavored filtered cigars
- Unflavored Filtered Cigars (Experimental): Half of the group will be randomized to start with unflavored FCs at the second visit and cross over to flavored FCs at the third visit. FCs will be Cheyenne filtered cigars.
  Interventions: Other: Unflavored filtered cigars

INTERVENTIONS:
Other: Flavored filtered cigars — Flavored and unflavored Cheyenne filtered cigars that are currently available in the marketplace for purchase
  Arms: Flavored Filtered Cigars
Other: Unflavored filtered cigars — Flavored and unflavored Cheyenne filtered cigars that are currently available in the marketplace for purchase
  Arms: Unflavored Filtered Cigars

SUMMARY:
The purpose of this study is to understand addiction to filtered cigars (FCs) compared to cigarettes in young adults, ages 21-34, who smoke both cigarettes and cigars. We are also looking to see if flavors, such as fruit or menthol, make FCs more addictive and if there are differences between men and women. Participants will receive 2 weeks supply of FCs, one week flavored and another week unflavored. You will be randomized (like flipping a coin) to which type of FC you will receive first. The study will:

* take about 3-4 hours of your time per week over 3-5 weeks.
* be conducted remotely by phone, video call, email, and mail.
* require a smart phone to answer 5 quick surveys a day
* you will need to answer 4 weekly surveys
* take part in a weekly video or phone call with research staff
* supply three saliva samples to be later tested for nicotine and other toxicants
* and use a device to measure your carbon monoxide levels four times a day.

You will be compensated for your time.

DETAILED DESCRIPTION:
The purpose of this remote study is to understand addiction to filtered cigars (FCs) compared to cigarettes in young adults, ages 21-34, who are dual users of cigarettes and cigars, if flavor, such as fruit or menthol, makes FCs more addictive, and if there are differences for men and women. The first hypothesis is that the potential for FCs to cause addiction will be lower than that of cigarettes but will increase as cigarette cost increases. Second, flavored FCs will be more addictive than unflavored FCs, and that the effect of flavored FCs on addiction will be greater in women than men. Last, participants will smoke more FCs and fewer cigarettes when given flavored compared to unflavored FCs. This study employs a crossover design (controlled for menthol status) in which 145 young adult dual users will be randomized to a flavored or unflavored FC that will be provided and then switch to the other type after 1 week. We will utilize the Cigarette Purchase Task, other standardized measures of dependence, and ecological momentary assessments to study the relationship between dependence indicators and smoking in the natural environment. Participation will take 3-4 hours of time per week over 3-5 weeks. Participants will be asked to complete brief surveys on their mobile phone 5 times a day, every day, weekly surveys about tobacco use, attitudes, and beliefs, and take part in a weekly video or phone call with research staff. They will need to use a carbon monoxide device we provide, four times a day, and provide 3 saliva samples that will later be analyzed for nicotine and other toxicants. All procedures will be conducted remotely by phone, computer, and mail.

ELIGIBILITY:
Inclusion Criteria:

* Current regular dual uses of filtered cigars and cigarillos (FCs) and cigarettes defined as; (a) report smoking cigarettes at least weekly in the past 30 days, (b) report smoking unaltered FC (without marijuana) at least weekly in the past 30 days; and (c)report cigarette and cigar use at their current rate (or more frequently) for ≥ 3 months.
* Able to read, speak, and understand English
* Age 21-34 years
* Stable residence (does not intend to move during the study period)
* Not intending to quit smoking during the study period
* Has a smart phone with a data plan (this study is being done remotely)
* Saliva cotinine level >30 ng/mL

Exclusion Criteria:

* Self-reported current pregnancy, currently trying to become pregnant, or breast-feeding
* Current use of nicotine replacement products or cessation products (e.g., bupropion) or plans to use in the next 3 weeks for the purposes of cessation.
* Diagnosed with or being treated for COPD, emphysema, and/or uncontrolled asthma as determined by research screening.
* Currently taking anti-hypertensive medications
* Currently has pneumonia, bronchitis, or COVID symptoms that has not yet resolved, or was hospitalized or visited the ER in the past 4 weeks for a respiratory-related illness that has not yet resolved (can be re-screened once resolved)
* Resident of Alaska, Hawaii, or Massachusetts

Ages: 21 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Change in demand elasticity for preferred flavored filtered cigars | 3-5 weeks
  It is measured by the Cigarette Purchase Task, which will be adapted to assess these products. It is the hypothetical consumption of flavored cigars at increasing prices.
Change in demand elasticity for preferred unflavored filtered cigars | 3-5 weeks
  It is measured by the Cigarette Purchase Task, which will be adapted to assess these products. It is the hypothetical consumption of unflavored cigars at increasing prices.
Change in cross price elasticity for filtered cigars and cigarettes | 3-5 weeks
  It is measured by the Cross-Price Purchase Task. It is the hypothetical consumption of flavored and unflavored filtered cigars as cigarette prices increase.

SECONDARY OUTCOMES:
Change in exhaled breath carbon monoxide (CO) level | 3-5 weeks
  Daily exhaled breath CO measured over the course of the study period

OTHER OUTCOMES:
Change in saliva cotinine levels | 3-5 weeks
  Saliva samples will be analyzed for cotinine levels
Change in number of flavored cigars, unflavored cigars, and cigarettes smoked per day | 3-5 weeks
  Participants will record tobacco use daily on their mobile phones using an app.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Mead-Morse, PhD,MHS, Principal Investigator — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
A verified database will be available once the main findings from the final dataset have been reported and accepted for publication. Information that does result from our analysis of the saliva samples will be available after publication of the findings. De-identified dataset will contain the data merged from all study visits. We will include with the data file proper documentation of all data (including definitions of variables and derived variables, frequencies, details about codes, etc.), and procedures used to collect the data, to ensure others can use the dataset and to prevent misuse, misinterpretation, and/or confusion. The database intended for public distribution will be free of identifiers that would permit linkages to individual research participants and variables that could lead to deductive disclosure of the identity of individual subjects.
Time Frame: In the final year of the Award after the dataset is finalized we will prepare a file in Excel and Stata that contains all study variables intended for use in presentations and publications.